CLINICAL TRIAL: NCT03818867
Title: Study Title: Emergency Cerclage in Twin Pregnancies at Imminent Risk of Preterm Birth: an Open-Label Randomised Controlled Trial
Brief Title: Emergency Cerclage in Twin Pregnancies at Imminent Risk of Preterm Birth: an Open-Label Randomised Controlled Trial
Acronym: ENCIRCLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17.004
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Preterm Birth; Twin Pregnancy With Antenatal Problem; Twin to Twin Transfusion Syndrome
Keywords: cervical cerclage; Preterm Birth; Twin pregnancy; Twin to Twin Transfusion Syndrome
MeSH Terms: conditions — Premature Birth; Fetofetal Transfusion | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage arm (Experimental): Pregnancies which had cervical cerclage inserted.
  Interventions: Procedure: Insertion of cervical cerclage
- No-cerclage arm (No Intervention): Pregnancies which did not have cervical cerclage inserted.

INTERVENTIONS:
Procedure: Insertion of cervical cerclage — insertion of a stitch around the neck of the womb in order to provide extra support.
  Other Names: cervical stitch
  Arms: Cerclage arm

SUMMARY:
Twin pregnancies are at an increased risk of early delivery. One of the reasons for this may be due to a weakened neck of the womb (cervix). There are 2 main ways to manage a weakened cervix in pregnancy. One option is to do nothing (conservative approach). The other is to strengthen the cervix with a stitch (cerclage) to provide extra support. There is no good quality convincing evidence to suggest which of these has better outcomes for mum and babies in twin pregnancies. This trial aims to determine whether securing the weakened cervix with a cerclage will help to prolong the pregnancy and prevent early delivery. Babies who are born early experience multiple complications including lung, brain and learning difficulties. Therefore, the study will also aim to determine whether prolonging the pregnancy by inserting the cerclage reduces the number of babies affected by these problems. In order to carry out a fair study we aim to perform what is known as a randomised controlled trial. We will include in the trial two major groups: (1) women pregnant with twins, who present with a weakened cervix and no signs of infection between 14 and 26 weeks of pregnancy. This will be diagnosed on an internal examination or ultrasound scan, and (2) women pregnant with identical twins complicated by twin-to-twin transfusion syndrome (TTTS) treated by Laser surgery between 16 and 26 weeks in whom a short cervix (<15mm) is identified. TTTS is rare but potentially devastating condition which occurs in about 10-15% of identical twin pregnancies. If left untreated, 80-90% of these babies will die. Overall, best first-line treatment of TTTS is laser surgery. Cervical length is a strong predictor of preterm delivery in these pregnancies.

Participants will be allocated randomly into the intervention (cerclage) or control (conservative) group. The procedure to insert the cerclage will be performed under an anaesthetic to minimise discomfort and you will be admitted for 2-3 days following the operation to ensure there are no complications or signs of labour. Women in both groups will be followed up in the same manner until they deliver and the pregnancy outcomes will be compared between the 2 groups to determine which management option is best.

DETAILED DESCRIPTION:
The study hypothesis is that the placement of an emergency cervical cerclage prolongs the pregnancy in (1) twin pregnancies with a dilated internal cervical os between 14+0 and 26+0 weeks, and (2) in monochorionic twin pregnancies complicated by TTTS treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (<15mm) is identified.

Study Design: Randomised controlled trial

Study population:

2 groups

* Twin pregnancies between 14 - 26 weeks' gestation presenting with an open cervix
* Monochorionic twin pregnancies complicated by twin-to-twin transfusion syndrome (TTTS) treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (<15mm) is identified

The primary outcome is time to delivery (from randomisation to birth). Secondary outcomes include gestation at delivery, preterm birth before 28, 32 and 34 weeks' gestation, birthweight, stillbirth, neonatal death, survival to discharge, days of admission to the neonatal intensive care unit, composite outcome of stillbirth, neonatal death, intraventricular haemorrhage, periventricular leukomalacia, respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy of prematurity, necrotising entercolitis, proven neonatal sepsis, or the need for ventilation, days of maternal admission for preterm labour and maternal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancies presenting with an open cervix between 14 and 26 weeks of gestation, OR
* Twin pregnancies complicated by TTTS treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (<15mm) is identified.
* Age >18 years
* Informed consent

Exclusion Criteria:

* Cervical dilatation ≥5cm
* Amniotic membranes prolapsed beyond external os into the vagina, unable to visualise cervical tissue
* Preterm premature rupture of the membranes (PPROM) at the time of diagnosis of dilated cervix
* Major fetal malformations unrelated to TTTS
* Intrauterine death of one or both fetuses
* Symptoms or signs of threatened imminent delivery, e.g. painful regular uterine contractions, active vaginal bleeding, history of ruptured membranes
* Suspected chorioamnionitis [based on maternal uterine tenderness, a temperature of 38°C or greater, significant leucocytosis (>15,000 x 106/L) or elevated C-reactive protein (>15 mg/L), or maternal tachycardia].
* Placenta praevia
* Monochorionic monoamniotic twin pregnancies
* Prophylactic cervical cerclage
* Women who are not able to give valid consent, e.g. unconscious or severely ill
* Mental health disorder which impairs the ability to give fully informed consent
* Women under the age of 18 years
* Higher order multiple pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to delivery (from randomisation to birth). | 2 weeks after expected date of birth
  Time between randomisation and delivery in days

SECONDARY OUTCOMES:
Gestation at delivery | 2 weeks after expected date of birth
  gestational age at delivery in weeks
Preterm birth before 28, 32 and 34 weeks' gestation | 2 weeks after expected date of birth
  the proportion of women giving birth before 28, 32 and 34 weeks
Birthweight | 42 days (28 days neonatal period+2 weeks postdates)
  birth weight in grams
Stillbirth | 42 days (28 days neonatal period+2 weeks postdates)
  death of the fetus (after 24 weeks) and before birth
Neonatal death | 42 days (28 days neonatal period+2 weeks postdates)
  the death of a baby within the first 28 days of life
Survival to discharge | 42 days (28 days neonatal period+2 weeks postdates)
  the proportion of the babies surviving until discharge from the hospital after birth
Days of admission to the neonatal intensive care unit | 42 days (28 days neonatal period+2 weeks postdates)
  Number of days the baby was admitted in the neonatal intensive care unit
Composite outcome | 42 days (28 days neonatal period+2 weeks postdates)
  An outcome which includes any of these outcomes (stillbirth, neonatal death, intraventricular haemorrhage, periventricular leukomalacia, respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy of prematurity, necrotising entercolitis, proven neonatal sepsis, or the need for ventilation)
Days of maternal admission for preterm labour | 2 weeks after expected date of birth
  Number of days the mother was admitted to the hospital because of preterm labour
Maternal morbidity (deﬁned as thromboembolic complications, chorioamnionitis, urinary tract infection treated with antibiotics, pneumonia, endometritis, eclampsia, HELLP syndrome, death, or any other significant morbidity) | 2 weeks after expected date of birth
  complications to the mother related to preterm labour or the insertion of the stitch

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khalil, Principal Investigator — St George's NHS Healthcare Trust
Locations (1):
- St George's Hospital, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03818867/Prot_SAP_000.pdf